CLINICAL TRIAL: NCT00320710
Title: A Prospective, Randomized, Double-blind, Stratified, Multi-center, 2-arm Trial of the Continued Efficacy and Safety of Zoledronic Acid (Every 4 Weeks vs. Every 12 Weeks) in in the 2nd Year of Treatment in Patients With Documented Bone Metastases From Breast Cancer
Brief Title: Continued Efficacy and Safety of Zoledronic Acid (q 4 Wks vs. q 12 Wks) in the 2nd Year of Treatment in Patients With Bone Metastases From Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CZOL446E2352
Record Dates: First submitted 2006-04-28; First posted 2006-05-03 (Estimated); Results first posted 2014-08-04 (Estimated); Last update posted 2014-08-22 (Estimated); Status verified 2014-08

CONDITIONS: Breast Cancer
Keywords: Breast cancer; zoledronic acid; bone metastases
MeSH Terms: conditions — Breast Neoplasms | interventions — Zoledronic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Zoledronic acid every (q) 4 weeks (Experimental): Participants received 4mg of zoledronic acid intravenously (IV) infusion q 4 weeks.
  Interventions: Drug: Zoledronic acid
- Zoledronic acid q 12 weeks (Experimental): Participants received 4 mg zoledronic acid IV q 12 weeks and received placebo to Zometa IV at the 4 week intervals between the q 12 week zoledronic acid infusions in order to maintain the blind.
  Interventions: Drug: Zoledronic acid; Drug: Placebo
- Placebo / zoledronic acid (Experimental): Participants randomized to this arm received placebo but the arm was later dropped and participants in this arm were swithced to the zoledronic acid q 4 weeks according to a study amendment.
  Interventions: Drug: Zoledronic acid; Drug: Placebo

INTERVENTIONS:
Drug: Zoledronic acid — 4mg IV
  Other Names: Zoledronate; ZOL446; Zometa
Drug: Placebo — Placebo to zoledronic acid
  Arms: Placebo / zoledronic acid; Zoledronic acid q 12 weeks

SUMMARY:
Clinical trial in breast cancer patients with bone metastases pretreated for approximately 1 year with a standard zoledronic acid regimen. Looking at the continued effectiveness and safety of giving zoledronic acid every 4 weeks versus every 12 weeks given over 1 year. This study is prospective, double-blind, stratified, multi-center, and two-arm.

ELIGIBILITY:
Inclusion Criteria:

Female patients ≥ 18 years of age. Confirmed breast cancer with bone metastasis. Pretreated with Zometa®, or Aredia (pamidronate) or all sequential regimens of both, for a minimum of 9 doses;

Exclusion Criteria:

Abnormal kidney function determined by serum creatinine levels. Current active dental problems including: ongoing infection of the teeth or jawbone; current exposed bone in the mouth; and current or prior diagnosis of osteonecrosis of the jaw.

Recent (within 8 weeks) or planned dental or jaw surgery (e.g., extraction, implants).

Diagnosis of metabolic bone disease other than osteoporosis (e.g., Paget's disease of bone).

Known hypersensitivity to Zometa. Treatment with other investigational drugs within 30 days prior to randomization.

Other protocol-defined exclusion criteria may have applied.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 416 (Actual)
Dates: Start 2006-02; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (92):
- United States (92):
  - Providence Alaska Medical Center Cancer Research, Anchorage, Alaska
  - Heritage Physicians Group Oncology, Hot Springs, Arkansas
  - The Center for Chest Care, Springdale, Arkansas
  - Pacific Cancer Medical Center, Inc., Anaheim, California
  - South Bay Oncology Hematology Partners, Campbell, California
  - Bay Area Cancer Research, Concord, California
  - Pacific Coast Hem/Onc, Fountain Valley, California
  - Wilshire Oncology Medical Group, La Verne, California
  - Kenmar Research Institute, Los Angeles, California
  - North Valley Hematology/Oncology Providence Holy Cross Medical, Northridge, California
  - Medical Oncology Care Associates, Orange, California
  - Ventura County Hematology and Oncology, Oxnard, California
  - The Office of Dr. Swarna Chanduri, MD, Pomona, California
  - Access Clinical Research, Rancho Mirage, California
  - Cancer and Blood of the Desert, Rancho Mirage, California
  - University of California Davis Cancer Center, Sacramento, California
  - University of California at Los Angeles, Sylmar, California
  - Denver Health Medical Center CACZ885M2301, Denver, Colorado
  - Eastern Connecticut Hematology & Oncology Associates, Norwich, Connecticut
  - Georgetown University/Lombardi Cancer Center, Washington D.C., District of Columbia
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Baptist Cancer Center, Jacksonville, Florida
  - Pasco Hernando Oncology, New Port Richey, Florida
  - The Office of Dr. Elizabeth Tan-Chiu, MD PA, Planatation, Florida
  - Suburban Hematology-Oncology, Lawrenceville, Georgia
  - NorthwesternUniv.Med.School/Robert H. Lurie Comp.Cancer Ctr, Chicago, Illinois
  - Evanston Northwestern Healthcare Medical Group, Evanston, Illinois
  - Edward Cancer Center, Naperville, Illinois
  - Midwest Cancer Research Group, Skokie, Illinois
  - Investigative Clinical Research, Indianapolis, Indiana
  - Cancer Care Center, New Albany, Indiana
  - Associated Physicians & Surgeons Clinic, Terre Haute, Indiana
  - Medical Associates Clinic, PC, Dubuque, Iowa
  - University of Iowa Health Care, Iowa City, Iowa
  - Siouxland Hematology-Oncology Associates LLP, Sioux City, Iowa
  - Cotton O'Neil Oncology Clinic, Topeka, Kansas
  - Cancer Center of Kansas, Witchita, Kansas
  - Kentucky Lung Clinic & Kentucky Sleep Clinic, Hazard, Kentucky
  - Lexington Oncology Associates, Lexington, Kentucky
  - Cabrini Center for Cancer Care, Alexandria, Louisiana
  - Southwest Oncology Associates Ltd., Lafayette, Louisiana
  - Greenbaum Cancer Center, Baltimore, Maryland
  - St. Agnes Hospital, Baltimore, Maryland
  - The Harry and Jeanette Weinberg Cancer Institute at Franklin, Baltimore, Maryland
  - Center for Cancer & Blood Disorders, Bethesda, Maryland
  - Frederick Memorial Hospital, Frederick, Maryland
  - Caritas Holy Family Hospital, Methuen, Massachusetts
  - University of Michigan Clinical Trials Office, Ann Arbor, Michigan
  - Wayne State University, Detroit, Michigan
  - Henry Ford Hospital Oncology, Detroit, Michigan
  - Oncology Care Associates, PLLC, Saint Joseph, Michigan
  - St. Luke's Hospital and Health Network, Duluth, Minnesota
  - Fairview Clinical Trial Services, Minneapolis, Minnesota
  - Univ. of Minnesota Cancer Center 420 Delaware St., Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center, Robbinsdale, Minnesota
  - Jackson Oncology Associates, Jackson, Mississippi
  - Capitol Comprehensive Cancer Care Clinic, Jefferson City, Missouri
  - The Center for Cancer Care and Research, St Louis, Missouri
  - Nebraska Hematology-Oncology PC, Lincoln, Nebraska
  - Nevada Cancer Centers 2851 North Tenaya Way, Las Vegas, Nevada
  - Center for Cancer and Hematologic Disease, Cherry Hill, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Somerset Hematology Oncology Associates, Somerset, New Jersey
  - Advanced Oncology Associates, Armonk, New York
  - Arena Oncology Associates, PC, Great Neck, New York
  - Benedictine Hospital, Kingston, New York
  - Beth Israel Medical Center, New York, New York
  - Columbia Presbyterian Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Jmaes P. Wilmot Cancer Center, Rochester, New York
  - Alamance Regional Medical Cancer Center, Burlington, North Carolina
  - Northeast Oncology Associates Suite 250, Concord, North Carolina
  - Barberton Citizens Hospital, Barberton, Ohio
  - Gabrail Cancer Center, Canton, Ohio
  - Ohio Cancer Specialists, Mansfield, Ohio
  - Hematology/Oncology Consultants Inc., West Worthington, Ohio
  - Trilogy Cancer Care, Wooster, Ohio
  - Bay Area Hospital - Pharmacy, Coos Bay, Oregon
  - The Corvallis Clinic, P.C., Corvallis, Oregon
  - Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Lancaster Cancer Center, Lancaster, Pennsylvania
  - U of Pittsburgh Cancer Institute Magee-Womens Hospital, Pittsburgh, Pennsylvania
  - Guthrie Cancer Center, Sayre, Pennsylvania
  - Mainline Oncology Hematology Assoc., Wynnewood, Pennsylvania
  - M. Francisco Gonzalez, MD., FACP, Columbia, South Carolina
  - Santee Hematology/Oncology, Sumter, South Carolina
  - MD Anderson Cancer Center/University of Texas 1155 Herman Pressler Street, Houston, Texas
  - Cancer Centers of South Texas, San Antonio, Texas
  - Providence Everett Medical Clinic, Everett, Washington
  - Seattle Cancer Care Alliance Seattle Cancer Care Alliance, Seattle, Washington
  - Rockwood Clinic Rockwood Clinic, PS, Spokane, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Hortobagyi GN, Van Poznak C, Harker WG, Gradishar WJ, Chew H, Dakhil SR, Haley BB, Sauter N, Mohanlal R, Zheng M, Lipton A. Continued Treatment Effect of Zoledronic Acid Dosing Every 12 vs 4 Weeks in Women With Breast Cancer Metastatic to Bone: The OPTIMIZE-2 Randomized Clinical Trial. JAMA Oncol. 2017 Jul 1;3(7):906-912. doi: 10.1001/jamaoncol.2016.6316. PMID 28125763
- See also: Visit NovartisClinicalTrials.com: Pre-qualify for a trial, and view a list of trials and participating study centers. — http://www.novartisclinicaltrials.com/webapp/etrials/searchTrial.do?trialID=513

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The initial study design contained 3 arms: zoledronic acid q4 weeks, zoledronic acid q12 weeks and placebo q4 weeks. Due to a study amendment, the placebo arm was discontinued and participants in this treatment group were switched to the zoledronic acid q4 week group. These participants were not included in the efficacy analysis.
Groups:
- Placebo / Zoledronic Acid: Participants randomized to this arm received placebo but the arm was later dropped and participants in this arm were later switched to the zoledronic acid q 4 weeks according to a study amendment.
Period: Overall Study
Arm/Group | Zoledronic Acid Every (q) 4 Weeks | Zoledronic Acid q 12 Weeks | Placebo / Zoledronic Acid
Started | 200 | 203 | 13
Treated (Safety Set) | 198 | 202 | 13
Completed | 106 | 127 | 8
Not Completed | 94 | 76 | 5
Not completed — Disease progression | 24 | 19 | 2
Not completed — Death | 10 | 7 | 1
Not completed — Administrative problems | 1 | 2 | 0
Not completed — Withdrawal by Subject | 20 | 26 | 1
Not completed — Protocol Violation | 6 | 5 | 0
Not completed — Abnormal test procedure result(s) | 2 | 0 | 0
Not completed — Abnormal laboratory value(s) | 12 | 3 | 0
Not completed — Adverse Event | 18 | 14 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zoledronic Acid Every (q) 4 Weeks | Zoledronic Acid q 12 Weeks | Placebo / Zoledronic Acid | Total
Number analyzed (Participants) | 200 | 203 | 13 | 416
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.2 (11.10) | 58.6 (11.15) | 60.8 (12.19) | 58.9 (11.14)
Sex/Gender, Customized [Number; unit: participants] — All participants were female.
  participants | 200 | 203 | 13 | 416

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Who Experienced at Least One Skeletal Related Event (SRE)
Description: An SRE was defined as a pathologic fracture (vertebral and non-vertebral), spinal cord compression, radiation to bone or surgery to bone.
Time Frame: 52 weeks
Population: The population included participants who were in the zoledronic acid q4 weeks and zoledronic acid q12 weeks treatment groups.
Measure: Number; unit: Percentage of participants
Arm/Group | Zoledronic Acid Every (q) 4 Weeks | Zoledronic Acid q 12 Weeks
Number analyzed (Participants) | 200 | 203
Percentage of participants | 22 | 23.2

2. Secondary Outcome: Time to First SRE
Description: An SRE was defined as a pathologic bone fracture (vertebral and non-vertebral), spinal cord compression, radiation to bone, or surgery to bone. The time to first individual SRE was defined as the date of randomization to the date of first occurrence of any SRE.
Time Frame: 52 weeks
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Zoledronic Acid Every (q) 4 Weeks | Zoledronic Acid q 12 Weeks
Number analyzed (Participants) | 200 | 203
Days | NA [NA to NA] — The median was not estimable because there were too few events to calculate the median. | NA [NA to NA] — The median was not estimable because there were too few events to calculate the median.

3. Secondary Outcome: Time to First Individual Type of SRE
Description: Types of SREs analyzed were pathologic fractures (vertebral and non-vertebral), spinal cord compression, radiation to bone and surgery to bone. The time to first indvidual SRE was defined as the date of randomization to the date of the first occurrence of any individual SRE.
Time Frame: 52 weeks
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Zoledronic Acid Every (q) 4 Weeks | Zoledronic Acid q 12 Weeks
Number analyzed (Participants) | 200 | 203
Weeks
  Vertebral pathologic fractures | NA [NA to NA] — The median was not estimable because too few events occurred to calculate the median. | NA [NA to NA] — The median was not estimable because too few events occurred to calculate the median.
  Non-vertebral pathologic fractures | NA [NA to NA] — The median was not estimable because too few events occurred to calculate the median. | NA [NA to NA] — The median was not estimable because too few events occurred to calculate the median.
  Spinal cord compression | NA [NA to NA] — The median was not estimable because too few events occurred to calculate the median. | NA [NA to NA] — The median was not estimable because too few events occurred to calculate the median.
  Radiation to bone | NA [NA to NA] — The median was not estimable because too few events occurred to calculate the median. | NA [NA to NA] — The median was not estimable because too few events occurred to calculate the median.
  Surgery to bone | NA [NA to NA] — The median was not estimable because too few events occurred to calculate the median. | NA [NA to NA] — The median was not estimable because too few events occurred to calculate the median.

4. Secondary Outcome: Change From Baseline in Mean Composite Brief Pain Inventory (BPI) Score
Description: Participants completed a BPI short form which is a 9 item self-administered questionnaire used to evaluate the severity of a participant's pain and the impact of this pain on the participant's daily functioning. The participant rates his or her worst, least, average, and current pain intensity, lists current treatments and perceived effectiveness, and rates the degree that pain interferes with general activity, mood, walking ability, normal work, relations with other persons, sleep, and enjoyment of life on a 10 point scale. The BPI composite score, which was calculated as the average of items 3, 4, 5 and 6 (worst pain, least pain, average pain and pain right now), ranged from 0 (best possible outcome, no pain) to 10 (worst possible outcome, pain as bad as you can imagine). A positive change from baseline indicates worsening.
Time Frame: baseline, 52 weeks
Population: The population included participants who were in the zoledronic acid q4 weeks and zoledronic acid q12 weeks treatment groups and had both baseline and week 52 values.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Zoledronic Acid Every (q) 4 Weeks | Zoledronic Acid q 12 Weeks
Number analyzed (Participants) | 89 | 100
scores on a scale | 0.24 (1.976) | 0.31 (2.099)

5. Secondary Outcome: Change From Baseline in Mean Analgesic Score
Description: The analgesic score indicates the types of pain medication used. The scores range as follows: 0 = none medication; 1 = minor analgesics (aspirin, NSAID, acetaminophen, propoxyphene, etc.); 2 = Tranquilizers, antidepressants, muscle relaxants, and steroids; 3 = Mild narcotics (oxycodone, meperidine, codeine, etc.); and 4 = Strong narcotics (morphine, hydromorphone, etc.). A positive change from baseline indicates worsening.
Time Frame: baseline, 52 weeks
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Zoledronic Acid Every (q) 4 Weeks | Zoledronic Acid q 12 Weeks
Number analyzed (Participants) | 94 | 104
score | 0.5 (1.28) | 0.5 (1.13)

6. Secondary Outcome: Change From Baseline in Urinary N-telopeptide / Creatinine Ratio
Description: Urine samples were collected to obtain n-telopeptide and creatinine values.
Time Frame: baseline, 48 weeks
Population: The population included participants who were in the zoledronic acid q4 weeks and zoledronic acid q12 weeks treatment groups and had both baseline and week 48 values.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Zoledronic Acid Every (q) 4 Weeks | Zoledronic Acid q 12 Weeks
Number analyzed (Participants) | 106 | 119
ratio | 10.612 (40.4073) | 14.697 (57.7315)

7. Secondary Outcome: Change From Baseline in Serum Bone Specific Alkaline Phosphatase
Description: Serum samples were collected to obtain bone specific alkaline phosphatase values.
Time Frame: baseline, 48 weeks
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mcg/L
Arm/Group | Zoledronic Acid Every (q) 4 Weeks | Zoledronic Acid q 12 Weeks
Number analyzed (Participants) | 93 | 105
mcg/L | 0.797 (27.8800) | 4.514 (12.4509)

8. Secondary Outcome: Skeletal Morbidity Rate
Description: An SMR for a patient was defined as the "number of occurrences" of any (or a particular) SRE allowing for only 1 event in any 3-week interval, divided by the "time at risk" in years. The "number of occurrences" and the "time at risk" were counts of SRE and the time from the randomization date. Counting began from randomization in the way that every counted event was followed by a 20-day period during which no SRE was counted, nor was the time counted as "at risk". For example, if a patient had 1 SRE during the study, the "time at risk" was calculated as the total number of days in the study minus the 20-day follow-up period for that SRE. If a patient had no SRE events, the entire study period was counted as "time at risk". This SMR calculation method had the advantage of avoiding multiple counts of possibly interdependent SREs (e.g. having 1 fracture increases the probability of having a subsequent SRE).
Time Frame: 52 weeks
Population: This population included all participants who were in the zoledronic acid q 4 weeks and zoledronic acid q 12 weeks treatment groups.
Measure: Mean (Standard Deviation); unit: Number of events per year
Arm/Group | Zoledronic Acid Every (q) 4 Weeks | Zoledronic Acid q 12 Weeks
Number analyzed (Participants) | 200 | 203
Number of events per year | 0.46 (1.063) | 0.50 (1.500)

ADVERSE EVENTS:
Arm/Group | Zoledronic Acid Every (q) 4 Weeks | Zoledronic Acid q 12 Weeks | Placebo / Zoledronic Acid
Serious Adverse Events (participants affected / at risk) | 50/198 | 51/202 | 3/13
Other Adverse Events (participants affected / at risk) | 182/198 | 185/202 | 12/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Zoledronic Acid Every (q) 4 Weeks (N=198) | Zoledronic Acid q 12 Weeks (N=202) | Placebo / Zoledronic Acid (N=13)
Anaemia (Blood and lymphatic system disorders) | 1 | 3 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 2 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 2 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0
Arteriovenous malformation (Congenital, familial and genetic disorders) | 0 | 1 | 0
Hypercalcaemia of malignancy (Endocrine disorders) | 1 | 0 | 0
Eye swelling (Eye disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 5 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 3 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 0
Megacolon (Gastrointestinal disorders) | 1 | 0 | 0
Mesenteric vein thrombosis (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 2 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 1 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0
Oral disorder (Gastrointestinal disorders) | 0 | 1 | 0
Varices oesophageal (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 2 | 0
Asthenia (General disorders) | 1 | 1 | 0
Disease progression (General disorders) | 1 | 0 | 0
Drug withdrawal syndrome (General disorders) | 0 | 1 | 0
Fibrosis (General disorders) | 0 | 1 | 0
General physical health deterioration (General disorders) | 2 | 2 | 0
Generalised oedema (General disorders) | 1 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 1 | 1
Oedema peripheral (General disorders) | 0 | 1 | 0
Pain (General disorders) | 2 | 0 | 0
Perforated ulcer (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Biliary dilatation (Hepatobiliary disorders) | 0 | 1 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1 | 0
Escherichia sepsis (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 4 | 1 | 0
Sepsis (Infections and infestations) | 2 | 0 | 0
Septic shock (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Comminuted fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 3 | 0
Hepatic enzyme increased (Investigations) | 1 | 0 | 0
Troponin increased (Investigations) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 4 | 4 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 2 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Brain mass (Nervous system disorders) | 0 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 0
Coma (Nervous system disorders) | 1 | 0 | 0
Convulsion (Nervous system disorders) | 1 | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0 | 0
Encephalopathy (Nervous system disorders) | 1 | 0 | 0
Hemiparesis (Nervous system disorders) | 1 | 0 | 0
Hepatic encephalopathy (Nervous system disorders) | 1 | 0 | 0
Hydrocephalus (Nervous system disorders) | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0
Somnolence (Nervous system disorders) | 1 | 1 | 0
Spinal cord compression (Nervous system disorders) | 0 | 1 | 0
Vasogenic cerebral oedema (Nervous system disorders) | 0 | 1 | 0
Acute psychosis (Psychiatric disorders) | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 2 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 2 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 2 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Zoledronic Acid Every (q) 4 Weeks (N=198) | Zoledronic Acid q 12 Weeks (N=202) | Placebo / Zoledronic Acid (N=13)
Anaemia (Blood and lymphatic system disorders) | 25 | 32 | 1
Leukopenia (Blood and lymphatic system disorders) | 9 | 11 | 0
Neutropenia (Blood and lymphatic system disorders) | 12 | 21 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 6 | 1
Palpitations (Cardiac disorders) | 2 | 1 | 1
Pericardial effusion (Cardiac disorders) | 2 | 1 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 1
Vision blurred (Eye disorders) | 4 | 4 | 1
Abdominal pain (Gastrointestinal disorders) | 20 | 15 | 2
Abdominal pain upper (Gastrointestinal disorders) | 12 | 4 | 0
Constipation (Gastrointestinal disorders) | 43 | 35 | 1
Diarrhoea (Gastrointestinal disorders) | 39 | 35 | 2
Dry mouth (Gastrointestinal disorders) | 11 | 5 | 0
Dyspepsia (Gastrointestinal disorders) | 8 | 16 | 1
Dysphagia (Gastrointestinal disorders) | 8 | 7 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 8 | 11 | 1
Nausea (Gastrointestinal disorders) | 57 | 51 | 3
Oesophagitis (Gastrointestinal disorders) | 1 | 4 | 1
Oral disorder (Gastrointestinal disorders) | 2 | 1 | 1
Stomatitis (Gastrointestinal disorders) | 20 | 8 | 2
Swollen tongue (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 30 | 33 | 4
Asthenia (General disorders) | 12 | 15 | 1
Chills (General disorders) | 10 | 9 | 0
Fatigue (General disorders) | 60 | 68 | 3
Oedema (General disorders) | 3 | 3 | 1
Oedema peripheral (General disorders) | 26 | 26 | 3
Pain (General disorders) | 15 | 11 | 0
Pyrexia (General disorders) | 18 | 21 | 1
Nasopharyngitis (Infections and infestations) | 14 | 13 | 0
Oral herpes (Infections and infestations) | 3 | 1 | 2
Sinusitis (Infections and infestations) | 11 | 18 | 2
Tooth infection (Infections and infestations) | 3 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 18 | 23 | 1
Urinary tract infection (Infections and infestations) | 15 | 23 | 2
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 3 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 1 | 2 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 2 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 2 | 4 | 1
Alanine aminotransferase increased (Investigations) | 8 | 9 | 1
Aspartate aminotransferase increased (Investigations) | 13 | 9 | 2
Blood albumin decreased (Investigations) | 2 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 15 | 9 | 2
Blood bilirubin increased (Investigations) | 3 | 2 | 1
Blood cholesterol increased (Investigations) | 0 | 0 | 1
Blood creatinine increased (Investigations) | 10 | 4 | 2
Blood glucose increased (Investigations) | 3 | 2 | 1
Blood lactate dehydrogenase increased (Investigations) | 7 | 7 | 1
Blood potassium decreased (Investigations) | 3 | 3 | 2
Blood urea increased (Investigations) | 3 | 1 | 1
Liver function test abnormal (Investigations) | 3 | 2 | 1
Red blood cell count decreased (Investigations) | 1 | 1 | 1
Serum ferritin decreased (Investigations) | 0 | 0 | 1
Weight decreased (Investigations) | 15 | 18 | 1
Weight increased (Investigations) | 4 | 4 | 1
Decreased appetite (Metabolism and nutrition disorders) | 31 | 27 | 0
Dehydration (Metabolism and nutrition disorders) | 8 | 9 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 3 | 3 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 2 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 19 | 20 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 65 | 56 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 52 | 38 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 18 | 20 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 15 | 18 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 | 6 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 29 | 25 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 32 | 30 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 14 | 15 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 8 | 12 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 49 | 48 | 3
Balance disorder (Nervous system disorders) | 6 | 5 | 1
Dizziness (Nervous system disorders) | 24 | 18 | 1
Headache (Nervous system disorders) | 33 | 34 | 1
Hypersomnia (Nervous system disorders) | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 11 | 12 | 1
Migraine (Nervous system disorders) | 0 | 1 | 1
Neuralgia (Nervous system disorders) | 1 | 4 | 1
Neuropathy peripheral (Nervous system disorders) | 20 | 21 | 3
Paraesthesia (Nervous system disorders) | 13 | 12 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 9 | 7 | 1
Restless legs syndrome (Nervous system disorders) | 1 | 0 | 1
Somnolence (Nervous system disorders) | 2 | 3 | 1
Anxiety (Psychiatric disorders) | 15 | 11 | 2
Depression (Psychiatric disorders) | 13 | 8 | 0
Insomnia (Psychiatric disorders) | 18 | 19 | 2
Pollakiuria (Renal and urinary disorders) | 1 | 4 | 1
Vaginal discharge (Reproductive system and breast disorders) | 0 | 2 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 22 | 27 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 32 | 26 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 12 | 11 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10 | 8 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 9 | 13 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 11 | 10 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 6 | 6 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 6 | 14 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 11 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 18 | 14 | 1
Aortic aneurysm (Vascular disorders) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 3 | 1 | 1
Hot flush (Vascular disorders) | 13 | 11 | 1
Hypertension (Vascular disorders) | 11 | 12 | 2
Lymphoedema (Vascular disorders) | 6 | 8 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.